CLINICAL TRIAL: NCT05147337
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2511 in Healthy Adult and Elderly Subjects
Brief Title: A Study to Assess the Safety and Tolerability of E2511 in Healthy Adult and Elderly Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E2511-A001-005
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: E2511; Healthy Participants; Elderly Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: E2511 10 mg or Placebo (Experimental): Non-Japanese adult (greater than or equal to [>=] 18 years and less than [<] 55 years old) participants will receive 10 milligram (mg) E2511 or E2511 matched placebo, tablets, orally, once daily from Day 1 to Day 14.
  Interventions: Drug: E2511; Drug: Placebo
- Cohort 2: E2511 20 mg or Placebo (Experimental): Non-Japanese adult participants will receive 20 mg E2511 or E2511 matched placebo, tablets, orally, once daily from Day 1 to Day 14.
  Interventions: Drug: E2511; Drug: Placebo
- Cohort 3: E2511 40 mg or Placebo (Experimental): Non-Japanese adult participants will receive 40 mg E2511 or E2511 matched placebo, tablets, orally, once daily from Day 1 to Day 14.
  Interventions: Drug: E2511; Drug: Placebo
- Cohort 4: E2511 80 mg or Placebo (Experimental): Non-Japanese adult participants will receive 80 mg E2511 or E2511 matched placebo, tablets, orally, once daily from Day 1 to Day 14.
  Interventions: Drug: E2511; Drug: Placebo
- Cohort 5: E2511 20 mg or Placebo (Experimental): Japanese adult (>=20 years and <55 years old) participants will receive 20 mg E2511 or E2511 matched placebo, tablets, orally, once daily from Day 1 to Day 14.
  Interventions: Drug: E2511; Drug: Placebo
- Cohort 6: E2511 40 mg or Placebo (Experimental): Japanese adult participants will receive 40 mg E2511 or E2511 matched placebo, tablets, orally, once daily from Day 1 to Day 14.
  Interventions: Drug: E2511; Drug: Placebo
- Cohort 7: E2511 80 mg or Placebo (Experimental): Japanese adult participants will receive 80 mg E2511 or E2511 matched placebo, tablets, orally, once daily from Day 1 to Day 14.
  Interventions: Drug: E2511; Drug: Placebo
- Cohort 8: E2511 40 mg or Placebo (Experimental): Non-Japanese older (>=55 years and less than or equal to [<=] 85 years old) participants will receive 40 mg E2511 or E2511 matched placebo, tablets, orally, once daily from Day 1 to Day 14.
  Interventions: Drug: E2511; Drug: Placebo

INTERVENTIONS:
Drug: E2511 — E2511 tablets.
Drug: Placebo — E2511 matched placebo tablets.

SUMMARY:
The primary objective of this study is to evaluate the safety, tolerability, and plasma pharmacokinetic (PK) of E2511 following multiple oral doses in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, male, or female, non-Japanese participants age >=18 years and <55 years old (Cohorts 1 to 4) or age >=55 years and <=85 years old (Cohort 8); or Japanese participants age >=20 years and <55 years old (Cohorts 5 to 7) at the time of informed consent
2. Japanese participants must also satisfy the following requirements:

   * Must have been born in Japan of Japanese parents and Japanese grandparents
   * Must have lived no more than 5 years outside of Japan
   * Must not have changed their lifestyle or habits, including diet, while living outside of Japan
3. Weight of at least 50 kilogram (kg) and body mass index (BMI) >=18 and <30 kilogram per square meter (kg/m^2) (Cohorts 1 to 7) or BMI >=18 and <32 kg/m^2 (Cohort 8) at Screening

Exclusion Criteria:

1. Females who are breastfeeding or pregnant at Screening or Baseline
2. Females of childbearing potential who:

   * Within 28 days before study entry, did not use a highly effective method of contraception
   * Do not agree to use a highly effective method of contraception throughout the entire study period and for 28 days after study drug discontinuation.
3. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
4. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
5. Evidence of disease within 4 weeks before dosing related to chronic headaches, migraines, joint pain, or other disorders or disease resulting in chronic or intermittent pain
6. Any personal or family history of seizures (including febrile seizures) or diagnosis of epilepsy or episode of unexplained loss of consciousness
7. Any history of neurological or other medical conditions which in the opinion of the investigator has the potential to reduce seizure threshold
8. Any history of gastrointestinal surgery that may affect PK profiles of E2511, example, hepatectomy, nephrectomy, digestive organ resection at Screening
9. Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment at Screening or Baseline
10. A prolonged QT/QT interval corrected for heart rate (QTc) interval or a prolonged QT/QTc interval (QT interval corrected for heart rate using Fridericia's formula [QTcF] greater than [>] 450 milliseconds [ms]). A history of risk factors for torsade de pointes
11. HR <50 or more than 100 beats per minute at Screening or Baseline (Cohorts 1 through 7); or HR <55 or more than 100 beats per minute at Screening or Baseline (Cohort 8) NOTE: At Baseline, HR must meet the above criteria on 3 assessments (each separated by 15 minutes) to ensure eligibility
12. Left bundle branch block
13. History of myocardial infarction or active ischemic heart disease
14. History of clinically significant arrhythmia or uncontrolled arrhythmia
15. Any lifetime history of suicidal ideation or any lifetime history of suicidal behavior as indicated by the C-SSRS
16. Any lifetime history of psychiatric disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From Screening up to 14 days after the last dose of study drug (up to 56 days)
Number of Participants With Serious Adverse Events (SAEs) | From Screening up to 14 days after the last dose of study drug (up to 56 days)
Number of Participants With Clinically Significant Abnormal Laboratory Values | From Screening up to 14 days after the last dose of study drug (up to 56 days)
Number of Participants With Clinically Significant Abnormal Vital Signs Values | From Screening up to 14 days after the last dose of study drug (up to 56 days)
Number of Participants With Clinically Significant Abnormal Electrocardiograms (ECGs) Findings | From Screening up to 14 days after the last dose of study drug (up to 56 days)
Number of Participants With Clinically Significant Abnormal Ambulatory Blood Pressure | From Screening up to 14 days after the last dose of study drug (up to 56 days)
Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-suicide Severity Rating Scale (C-SSRS) | From Screening up to 14 days after the last dose of study drug (up to 56 days)
  The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess any suicidality, suicidal behavior, or suicidal ideation. Any suicidality is emergence of any suicidal ideation or suicidal behavior. Any suicidal behavior is indicated when response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation is indicated when response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide.
Number of Participants With Clinically Significant Abnormal Physical Examination Findings | From Screening up to 14 days after the last dose of study drug (up to 56 days)
Number of Participants With Clinically Significant Abnormal Neurological Examination Findings | From Screening up to 14 days after the last dose of study drug (up to 56 days)
Number of Participants With Clinically Significant Abnormal Electroencephalogram (EEG) Findings | From Screening up to 14 days after the last dose of study drug (up to 56 days)
Cmax: Maximum Observed Plasma Concentration for E2511 | Day 1: pre-dose up to 24 hours post-dose
Css,max: Maximum Observed Plasma Concentration at Steady State for E2511 | Day 14: pre-dose up to 24 hours post-dose
tmax: Time to Reach Maximum Observed Plasma Concentration (Cmax) for E2511 | Day 1: pre-dose up to 24 hours post-dose
tss,max: Time to Reach Maximum Observed Plasma Concentration (Cmax) at Steady State for E2511 | Day 14: pre-dose up to 24 hours post-dose
Css,av: Average Steady State Plasma Concentration for E2511 | Day 14: pre-dose up to 24 hours post-dose
AUC(0-t): Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration for E2511 | Day 1: pre-dose up to 24 hours post-dose; Day 14: pre-dose up to 24 hours post-dose
AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time Zero to Infinite for E2511 | Day 1: pre-dose up to 24 hours post-dose
AUC(0-24h): Area Under the Plasma Concentration-time Curve From Time Zero to 24 hours Post-dose for E2511 | Day 1: pre-dose up to 24 hours post-dose; Day 14: pre-dose up to 24 hours post-dose
t1/2: Terminal Elimination Phase Half-life for E2511 | Day 1: pre-dose up to 24 hours post-dose; Day 14: pre-dose up to 24 hours post-dose
PTF: Peak-trough Fluctuation for E2511 | Day 14: pre-dose up to 24 hours post-dose
CL/F: Apparent Total Clearance for E2511 | Day 1: pre-dose up to 24 hours post-dose
CLss/F: Apparent Total Clearance at Steady State for E2511 | Day 14: pre-dose up to 24 hours post-dose
Vz/F: Apparent Volume of Distribution at Terminal Phase for E2511 | Day 1: pre-dose up to 24 hours post-dose; Day 14: pre-dose up to 24 hours post-dose
Rac: Accumulation Ratio for E2511 Based on Cmax and AUC | Day 14: pre-dose up to 24 hours post-dose
Rss: Accumulation Ratio for E2511 Based on Time and Concentration | Day 14: pre-dose up to 24 hours post-dose

SECONDARY OUTCOMES:
Change From Baseline in the Concentration of Acetylcholine (ACh) in Cerebrospinal Fluid (CSF) | Baseline, Day 13
Change From Baseline in Heart Rate (HR) | Baseline up to Day 15
Change From Baseline in PR Interval of the ECG (PR), QRS Interval of the ECG (QRS), and QT Interval Corrected for Heart Rate (QTc) of the ECG | Baseline up to Day 15
Placebo Corrected Change From Baseline in HR | Baseline up to Day 15
Placebo Corrected Change From Baseline in PR, QRS, and QTc Interval | Baseline up to Day 15
Number of Participants With Categorical Outliers for HR, PR, QRS and QTc Interval | Baseline up to Day 15
Number of Participants With Treatment-emergent T-wave and U-wave abnormalities | Baseline up to Day 15
Mean Change From Baseline in 24-hours Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) up to Day 15 | Up to Day 15
  The blood pressure (BP) will be evaluated by Ambulatory Blood Pressure Monitoring (ABPM) for all participants based on the measurement of BP recordings after every 24 hours.
Mean Change From Baseline in Day-time, Night-time, and Hourly SBP and DBP | Baseline up to Day 15
Mean Change From Baseline in Day-time, Night-time, and Hourly HR | Baseline up to Day 15
Mean Change From Baseline in Day-time, Night-time, and Hourly Mean Arterial Pressure (MAP) and Pulse Pressure (PP) | Baseline up to Day 15
Placebo Corrected Mean Change From Baseline in 24-hours SBP and DBP up to Day 15 | Up to Day 15
  The BP will be evaluated by ABPM for all participants based on the measurement of BP recordings after every 24 hours.
Placebo Corrected Mean Change From Baseline in Day-time, Night-time, and Hourly SBP and DBP | Baseline up to Day 15
Placebo Corrected Mean Change From Baseline in Day-time, Night-time, and Hourly HR | Baseline up to Day 15
Placebo Corrected Mean Change From Baseline in Day-time, Night-time, and Hourly MAP and PP | Baseline up to Day 15
Number of Participants With Categorical Outliers for SBP and DBP | Baseline up to Day 15
Geometric Mean Ratio of Cmax Between the Healthy Japanese and Non-japanese Participants for E2511 | Day 1: pre-dose up to 24 hours post-dose; Day 14: pre-dose up to 24 hours post-dose
Geometric Mean Ratio of AUC Between the Healthy Japanese and Non-japanese Participants for E2511 | Day 1: pre-dose up to 24 hours post-dose; Day 14: pre-dose up to 24 hours post-dose
Geometric Mean Ratio of Cmax Between the Younger Non-japanese (>=18 and <55 years) and older Non-japanese (>=55 to <=85 years) Participants for E2511 | Day 1: pre-dose up to 24 hours post-dose; Day 14: pre-dose up to 24 hours post-dose
Geometric Mean Ratio of AUC Between the Younger Non-japanese (>=18 and <55 years) and older Non-japanese (>=55 to <=85 years) Participants for E2511 | Day 1: pre-dose up to 24 hours post-dose; Day 14: pre-dose up to 24 hours post-dose
Geometric Mean Ratio Between the Non-japanese (>=18 and <55 years) and Elderly Non-japanese (>=65 to <=85 years) Participants for E2511 | Day 1: pre-dose up to 24 hours post-dose; Day 14: pre-dose up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- California Clinical Trials Medical Group, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.